CLINICAL TRIAL: NCT00448227
Title: A Multicenter, Open-label, Single-arm Study to Evaluate the Single-dose Pharmacokinetics, Acceptability and Safety of Famciclovir Oral Pediatric Formulation in Infants 1 Month to Less Than 1 Year of Age With Herpes Simplex Virus Infections
Brief Title: Pharmacokinetics, Acceptability and Safety of Famciclovir in Infants (1 Month to Less Than 12 Months) With Herpes Simplex Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFAM810B2301
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Herpes Simplex
Keywords: Infants, Herpes simplex infection
MeSH Terms: conditions — Herpes Simplex | interventions — Famciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Famciclovir (Experimental): Famciclovir was administered orally as a suspension in OraSweet® on Day 1. Patients received a single, individualized dose between 25-200 mg based on body weight.
  Interventions: Drug: famciclovir

INTERVENTIONS:
Drug: famciclovir — Administered orally as a single individualized dose between 25-200 mg based on body weight.
  Other Names: Famvir

SUMMARY:
This study will evaluate the acceptability and safety of famciclovir in infants with herpes simplex infection

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 1 month up to 1 year of age with herpes simplex infection

Exclusion Criteria:

* Patients with gestational age less than 32 weeks. Patients unable to swallow. Patients with history of malabsorption or previous gastrointestinal surgery.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis; Dr. Jeffery L. Blumer, Principal Investigator — University Hospital Cased Medical Center Rainbow Babies and Children's Hospital, Cleveland, OH
Locations (6):
- United States (6):
  - Pediatric Infectious Disease Of University of Alabama, Birmingham, Alabama
  - Children's Memorial Hospital Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Archana Chatterjee, Omaha, Nebraska
  - University Hospital Cased Medical Center Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Blumer J, Rodriguez A, Sanchez PJ, Sallas W, Kaiser G, Hamed K. Single-dose pharmacokinetics of famciclovir in infants and population pharmacokinetic analysis in infants and children. Antimicrob Agents Chemother. 2010 May;54(5):2032-41. doi: 10.1128/AAC.01508-09. Epub 2010 Feb 16. PMID 20160046
- See also: Related Info — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Famciclovir
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Famciclovir
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: months] | 4 (3.60)
Age, Customized [Number; unit: participants]
  1 to <3 months | 8
  3 to <6 months | 5
  6 to 12 months | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Single Dose - Tmax
Description: Measured by Tmax - The time after administration of a drug when the maximum plasma concentration is reached.
Time Frame: Plasma samples were collected at 0.5, 1, 4 and 6 hours after dosing.
Population: Analysis population included the intent-to-treat population, with the exception of one patient in the 1 to <3 months age group who did not have PK samples taken due to emesis reported after study medication administration.
Measure: Median (Full Range); unit: hours
Groups:
- Famciclovir: Infants 1 to <3 Months: Infants 1 to <3 months. Famciclovir was administered orally as a suspension in OraSweet® on Day 1. Patients received a single, individualized dose between 25-200 mg based on body weight.
- Famciclovir: Infants 3 to <6 Months: Infants 3 to <6 months. Famciclovir was administered orally as a suspension in OraSweet® on Day 1. Patients received a single, individualized dose between 25-200 mg based on body weight.
- Famciclovir: Infants 6 to 12 Months: Infants 6 to 12 months. Famciclovir was administered orally as a suspension in OraSweet® on Day 1. Patients received a single, individualized dose between 25-200 mg based on body weight.
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months
Number analyzed (Participants) | 7 | 5 | 5
hours | 1.00 [1.00 to 5.17] | 4 [1.00 to 4.17] | 1.02 [0.58 to 1.10]

2. Secondary Outcome: Safety Assessed by AEs, SAEs
Description: AEs and SAEs were collected during patient's stay in the clinic for PK sampling up to Hour 8, then at day 2 visit, 8 days(safety follow-up call) and 38 days (safety follow-up call) post dose.
Time Frame: 38 days
Reporting Status: Not Posted

3. Secondary Outcome: Safety Assessed by Labs
Description: Samples for safety labs were obtained at baseline and Day 2 visit and samples were analyzed by local accredited laboratory.
Time Frame: 2 days
Reporting Status: Not Posted

4. Secondary Outcome: Tolerability of of the Famciclovir Pediatric Formulation as Assessed by Study Personnel.
Description: Tolerability was assessed by the study personnel 30 minutes after dosing using the following scale:
  1. Significant emesis occurred,
  2. Infant spit out most of the dose ingesting less than half of what was administered,
  3. Infant spit out some of the dose, but ingested at least 50% of what was administered,
  4. Infant was able to ingest and retain the dose administered
Time Frame: 30 minutes after dosing
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months | Total
Number analyzed (Participants) | 8 | 5 | 5 | 18
Participants
  Significant emesis occurred | 1 | 0 | 0 | 1
  Spit out most of the dose, ingested less than half | 0 | 0 | 0 | 0
  Spit out some of the dose, ingested at least 50% | 0 | 0 | 0 | 0
  Able to ingest and retain dose | 7 | 5 | 5 | 17

5. Secondary Outcome: Acceptability of the Famciclovir Pediatric Formulation as Assessed by the Patient's Caregiver
Description: Assessed by the caregiver using a 5-point scale immediately after dosing:
  1. Very badly accepted/unacceptable: infant showed great displeasure, compromising use of formulation
  2. Badly but accepted: infant showed displeasure with dosing but could be coaxed to take complete dose
  3. Neither good nor bad: infant showed no apparent displeasure and with little effort was coaxed to take complete dose
  4. Well accepted: infant appeared to enjoy the formulation and with little coaxing ingested most of dose
  5. Very well accepted: infant appeared eager and ingested most of dose without special coaxing
Time Frame: Immediately after dosing
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months | Total
Number analyzed (Participants) | 8 | 5 | 5 | 18
Participants
  Very badly / unacceptable | 1 | 0 | 0 | 1
  Badly but accepted | 0 | 0 | 1 | 1
  Neither good nor bad | 0 | 2 | 1 | 3
  Well accepted | 2 | 0 | 2 | 4
  Very well accepted | 4 | 3 | 1 | 8

6. Primary Outcome: Pharmacokinetics of Single Dose - Cmax
Description: Measured by Cmax - The maximum plasma concentration of study medication
Time Frame: Plasma samples were collected at 0.5, 1, 4 and 6 hours after dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months
Number analyzed (Participants) | 7 | 5 | 5
μg/mL | 0.69 (0.41) | 0.74 (0.17) | 3.24 (1.01)

7. Primary Outcome: Pharmacokinetics of Single Dose - AUC(0-tlast)
Description: Measured by AUC(0-tlast) - Area under the plasma concentration time curve from time zero to the last quantifiable concentration-timepoint.
Time Frame: Plasma samples were collected at 0.5, 1, 4 and 6 hours after dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (μg/mL)•h
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months
Number analyzed (Participants) | 7 | 5 | 5
(μg/mL)•h | 2.09 (1.38) | 3.16 (0.68) | 8.68 (2.09)

8. Primary Outcome: Pharmacokinetics of Single Dose - AUC(0-6h)
Description: Measured by AUC(0-6h) - Area under the plasma concentration time curve from time zero up to 6 hours post dose (i.e. the time of the last sample).
Time Frame: Plasma samples were collected at 0.5, 1, 4 and 6 hours after dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (μg/mL)•h
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months
Number analyzed (Participants) | 7 | 5 | 5
(μg/mL)•h | 2.22 (1.23) | 3.16 (0.68) | 8.77 (2.14)

9. Secondary Outcome: Acceptability of the Famciclovir Pediatric Formulation as Assessed by Study Personnel
Description: Assessed by the study personnel using a 5-point scale after dosing:
  1. Very badly accepted/unacceptable: infant showed great displeasure, compromising use of formulation
  2. Badly but accepted: infant showed displeasure with dosing but could be coaxed to take complete dose
  3. Neither good nor bad: infant showed no apparent displeasure and with little effort was coaxed to take complete dose
  4. Well accepted: infant appeared to enjoy the formulation and with little coaxing ingested most of dose
  5. Very well accepted: infant appeared eager and ingested most of dose without special coaxing
Time Frame: Immediately after dosing
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Famciclovir: Infants 1 to <3 Months | Famciclovir: Infants 3 to <6 Months | Famciclovir: Infants 6 to 12 Months | Total
Number analyzed (Participants) | 8 | 5 | 5 | 18
Participants
  Very badly / unacceptable | 1 | 0 | 0 | 1
  Badly but accepted | 0 | 0 | 1 | 1
  Neither good nor bad | 0 | 2 | 2 | 4
  Well accepted | 2 | 0 | 1 | 3
  Very well accepted | 4 | 3 | 1 | 8

ADVERSE EVENTS:
Arm/Group | Famciclovir
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir (N=18)
Condition aggravated (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir (N=18)
Anaemia (Blood and lymphatic system disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 2
Oral candidiasis (Infections and infestations) | 1
Occult blood positive (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Encephalitis (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Condition aggravated (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is typically a disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.